CLINICAL TRIAL: NCT02686632
Title: Improving Practice Guidelines for the Treatment of Denture-related Erythematous Stomatitis: A Pragmatic International Multicenter Randomized Controlled Trial
Brief Title: The Effectiveness of Palatal Brushing on Denture Stomatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Elham Emami, Associate Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMD-UdeM-EE-2016a
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Denture Stomatitis
Keywords: Denture Stomatitis; Denture Erythematous Stomatitis; Prosthesis Stomatitis; Oral Candidiasis; Palatal inflammation
MeSH Terms: conditions — Stomatitis, Denture; Candidiasis, Oral

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palate Brushing (Experimental): In this group the intervention is "palatal brushing", performed by the participants following each meal for a period of 6 months. This will be performed using the provided toothbrush (device). The results will determine if brushing the palate in an efficient intervention for reducing the microbial count and inflammation associated with denture stomatitis.
  Interventions: Behavioral: Palatal brushing
- Regular Oral Hygiene (No Intervention): The participants in this study arm will not be prescribed or allocated any intervention. The participants will be asked to continue with the regular hygiene and denture maintenance practices for the duration of the trial.

INTERVENTIONS:
Behavioral: Palatal brushing — Brushing the palate as part of regular oral hygiene habits (behavior) among complete denture wearers.
  Arms: Palate Brushing

SUMMARY:
Denture stomatitis (DS) is an oral biofilm associated inflammatory disease of the palatal mucosa. It is the most prevalent oral disease and the main indicator of poor oral health among denture wearers, affecting one-third of all complete denture wearers.

The etiology of DS is multifactorial, with documented role of mechanical trauma, bacteria and fungi. Risk factors may include, poor oral hygiene and nocturnal use of dentures. However, the evidence is ambiguous, inconclusive and recurrence following routine antifungal therapy is common.

The proposed study is a phase II clinical trial to evaluate the efficacy of palatal brushing in reducing the colony forming unit (CFU) count and clinical inflammation. The assessment of change in CFU count and clinical inflammation will be carried out at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Wearing a maxillary and mandibular complete conventional denture
* Having moderate to severe signs of denture stomatitis according to Schwartz index
* Providing consent prior to study.

Exclusion Criteria:

* Oral mucosal lesions other than denture stomatitis.
* Systemic conditions which predispose to Candida specie infection such as uncontrolled diabetes and xerostomia.
* History of chemotherapy/radiotherapy.
* Used antibiotics, steroidal or antifungal agents in the 4 weeks prior to the study.
* Scheduled to replace existing dentures with new ones during the length of the trial.
* Already using palatal brushing as a routine oral hygiene procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Candida species colony forming units | Baseline to 6 months
  Palatal saliva (swab) and denture sonicate will be analysed for Candida species CFU count at baseline, 3 months and 6 months. The results will be presented as change in mean CFU count.

SECONDARY OUTCOMES:
Clinical Inflammation | Baseline to 6 months
  Change in clinical inflammation will be examined and recorded in both groups at baseline, 3 months and 6 months and presented as change in mean inflammation scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jainkittivong A, Aneksuk V, Langlais RP. Oral mucosal lesions in denture wearers. Gerodontology. 2010 Mar;27(1):26-32. doi: 10.1111/j.1741-2358.2009.00289.x. PMID 20461847
- [Background] Gendreau L, Loewy ZG. Epidemiology and etiology of denture stomatitis. J Prosthodont. 2011 Jun;20(4):251-60. doi: 10.1111/j.1532-849X.2011.00698.x. Epub 2011 Apr 4. PMID 21463383
- [Background] Slade GD, Akinkugbe AA, Sanders AE. Projections of U.S. Edentulism prevalence following 5 decades of decline. J Dent Res. 2014 Oct;93(10):959-65. doi: 10.1177/0022034514546165. Epub 2014 Aug 21. PMID 25146182
- [Background] de Oliveira CE, Gasparoto TH, Dionisio TJ, Porto VC, Vieira NA, Santos CF, Lara VS. Candida albicans and denture stomatitis: evaluation of its presence in the lesion, prosthesis, and blood. Int J Prosthodont. 2010 Mar-Apr;23(2):158-9. PMID 20305856
- [Background] Emami E, de Grandmont P, Rompre PH, Barbeau J, Pan S, Feine JS. Favoring trauma as an etiological factor in denture stomatitis. J Dent Res. 2008 May;87(5):440-4. doi: 10.1177/154405910808700505. PMID 18434573
- [Background] Cross LJ, Williams DW, Sweeney CP, Jackson MS, Lewis MA, Bagg J. Evaluation of the recurrence of denture stomatitis and Candida colonization in a small group of patients who received itraconazole. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Mar;97(3):351-8. doi: 10.1016/j.tripleo.2003.10.006. PMID 15024360
- [Derived] de Souza RF, Khiyani MF, Chaves CAL, Feine J, Barbeau J, Fuentes R, Borie E, Crizostomo LC, Silva-Lovato CH, Rompre P, Emami E. Improving practice guidelines for the treatment of denture-related erythematous stomatitis: a study protocol for a randomized controlled trial. Trials. 2017 May 5;18(1):211. doi: 10.1186/s13063-017-1947-y. PMID 28476133
- See also: Phase I clinical trial of the proposed study — http://www.ncbi.nlm.nih.gov/pubmed/25010873